CLINICAL TRIAL: NCT01740492
Title: Low Dose Ketamine for Management of Acute Severe Pain in the Emergency Department
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 298021
Record Dates: First submitted 2012-09-26; First posted 2012-12-04 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2012-09

CONDITIONS: Pain
Keywords: Ketamine; Acute pain; Pain control; Pain
MeSH Terms: conditions — Pain; Acute Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LDK1: Low dose Ketamine (0.15mg/kg) (Experimental): Participants randomized to the first group, LDK1, will receive an intravenous injection of low dose ketamine (0.15mg/kg).
  All participants, regardless of the group, will receive a dose of morphine(0.15mg/kg) at the same time the study drug is administered.
  Interventions: Drug: Ketamine 0.15mg/kg
- LDK2: Low dose Ketamine (0.3mg/kg) (Experimental): Participants randomized to the second group, LDK2, will receive an intravenous injection of low dose ketamine (0.3mg/kg).
  All participants, regardless of the group, will receive a dose of morphine(0.15mg/kg) at the same time the study drug is administered.
  Interventions: Drug: Ketamine 0.3mg/kg
- 0.9% Normal Saline (Placebo Comparator): This group will receive a placebo injection of 0.9% normal saline of a similar volume (0.05ml/kg)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine 0.15mg/kg — 0.15mg/kg ketamine delivered IV (in the vein) following clinician assessment in ER. Number of cycles: until discharge or 6 hours elapses.
  Other Names: Ketamine
  Arms: LDK1: Low dose Ketamine (0.15mg/kg)
Drug: Ketamine 0.3mg/kg — 0.3 mg/kg ketamine delivered IV (in the vein) following clinician assessment in ER. Number of cycles: until discharge or 6 hours elapses.
  Other Names: Ketamine
  Arms: LDK2: Low dose Ketamine (0.3mg/kg)
Other: Placebo — Placebo injection of 0.9% normal saline of a similar volume (0.05ml/kg)
  Arms: 0.9% Normal Saline

SUMMARY:
This study aims to address both the management and evaluation of pain. The primary aim of this study is to determine the efficacy of low dose ketamine in adults with moderate to severe pain in the emergency department as compared with parenteral opioids alone. Another aim is to examine the safety of low dose ketamine compared to opioids alone.

The investigators hypothesize that low dose ketamine will result in more effective pain control than morphine alone and will not be associated with an increase in adverse events.

DETAILED DESCRIPTION:
Management and assessment of pain in the Emergency Department (ED) can be challenging. Treatment of pain is most often accomplished by parenteral opioids analgesics. However, inadequate analgesia is often a problem when opioids alone are relied on for pain control. In the peri-operative setting ketamine has been used as an adjunct to opioids for acute pain. Ketamine may play a role in maximizing analgesia in the ED.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adults age 18-65
* Able to understand and give informed consent
* Comfortable with the experimental protocol as outlined to them by the research team
* Severe pain, pain score of at least 50/100 on Visual Analogue Scale (VAS) or 5/10 numerical ratings score
* Acute pain, pain duration < 7days
* Deemed by treating ED attending physician to require IV opioid analgesia
* ASA (American Society of Anesthesiologists) class I or II

Exclusion Criteria:

* Previously enrolled in the study
* Neurologic, respiratory, or hemodynamic compromise
* GCS (Glasgow Coma Scale) <15
* Pox <94%, RR <10, or RR >22
* SBP <90, SBP>180, or DBP >110
* Discretion of treating physician
* Pregnancy or breastfeeding
* Known or suspected allergy to ketamine or morphine
* Ketamine within 24 hours of presentation (prescription or illicit drugs)
* Conscious sedation in ED (per treating physician), includes ketamine (for non-study purposes)
* Known Renal (Cr>2.0) or Liver Failure
* Unstable psychiatric disease (as per treating physician)
* History of stroke
* History of cardiac disease
* Prior myocardial infarction; Angina (Stable or Unstable)
* Cardiac stents or bypass surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in reported pain score at 15 minutes, 30 minutes, and hourly for 6 hrs or until discharge | Between patient arrival and patient discharge
  At baseline, to assess our primary aim, efficacy of pain control, we will use patient reported pain scores and amount of rescue analgesia (parenteral morphine) received. Trained research assistants (RA) will ask participants to report their pains scores using a numerical pain rating scale (NPRS). The NPRS used will be a 0 to 10 rating scale: a rating of 0 corresponds to "no pain at all," whereas a rating of 10 is the "worst pain imaginable." Baseline NPRS will be measured after randomization, but just before administration of ketamine or placebo injection and morphine (Baseline). Repeat measurements will be taken at 15 minutes, 30 minutes, and hourly following treatment with the study drug, for 6hrs or until the patient leaves the ED. The amount of rescue analgesia will be recorded at each time point. The ED course will also be reviewed post hoc by the RAs and physician investigators to confirm analgesia received. The main outcome measure will be the change in pain score over time.

SECONDARY OUTCOMES:
Safety--Determine the incidence of adverse events associated with ketamine and morphine, versus morphine alone at 5 minutes, 30 minutes, and hourly up to 6 hours. | 15 minutes, 30 minutes, hourly up to 6 hours
  Adverse events will further be defined as Hypotension (SBP < 90), Hypertension (SBP >180, or Diastolic Blood Pressure >110), Presence of nausea/vomiting, presence of hallucinations, Respiratory depression (pOx<92%, Respirator Rate<12, EtCO2 >40), and need for naloxone. All patients will be monitored continuously with cardiac telemetry, pulse oximetry, and capnography following administration of the study drug. Level of sedation will be assessed using an adaptation of the Ramsay Scoring System and the Pasero Opioid Induced Sedation Scale. (Appendix 2) Further, the ED and inpatient course will be reviewed post hoc by the RAs and physician investigators who will record: Time to inpatient admission or discharge, inpatient length of stay, time to operative intervention, outcome of admission (i.e. discharge to home, SNF, rehab) and any morbidity and mortality suffered by the patient and medical complications (myocardial infarction, respiratory infection, etc…).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Beaudoin, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States